CLINICAL TRIAL: NCT05089929
Title: Endoscopic Esophageal Topography (Endoflip 2.0) Versus High-resolution Manometry (HRM) in Pre-operative Evaluation of GERD; a Non-inferiority Trial
Brief Title: Endoscopic Esophageal Topography (Endoflip 2.0) Versus High-resolution Manometry (HRM)
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Kelly Haisley, Assistant Professor, Ohio State University
Other Study IDs: 2020H0057
Record Dates: First submitted 2021-06-14; First posted 2021-10-22 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Endoflip 2.0: The investigators will perform FLIP topography (Endoflip 2.0) analysis on all patients undergoing routine evaluation for gastroesophageal reflux disease at the time of their pre-operative EGD.
  Interventions: Device: Endoflip 2.0; Procedure: High Resolution Manometry

INTERVENTIONS:
Device: Endoflip 2.0 — FLIP topography (Endoflip 2.0) analysis will be performed on all patients undergoing routine evaluation for gastroesophageal reflux disease at the time of their pre-operative EGD.
Procedure: High Resolution Manometry — All patients undergoing routine evaluation for gastroesophageal reflux disease will undergo high resolution manometry (HRM) testing.

SUMMARY:
The purpose of the study is to investigate the use of FLIP topography in patients undergoing evaluation for gastroesophageal reflux disease (GERD). This device allows the clinician to measure muscle activity in the esophagus during a routine upper endoscopy. The FLIP topography will be used to help detect movement disorders in the esophagus, and to examine differences in patient satisfaction between FLIP topography and the standard of care procedure, high resolution manometry (HRM).

DETAILED DESCRIPTION:
The goal of the proposed research is to evaluate the endoscopic esophageal functional luminal imaging probe (FLIP) with topography (Endoflip® 2.0, Medtronic, USA) as a pre-operative diagnostic test to rule out significant esophageal dysmotility in patients with gastroesophageal reflux disease (GERD). Currently, the gold standard for pre-operative motility assessment is high resolution manometry (HRM), a trans-nasal catheter test performed in an awake patient that can be quite uncomfortable, and some patients cannot tolerate.1 Conversely, Endoflip can provide similar data in a sedated patient at the time of upper endoscopy, limiting discomfort and streamlining workup. While Endoflip has been used as a complimentary tool for clinical decision making in major motility disorders, its evaluation as a potential stand-alone pre-operative test in the GERD population has been limited. However, if FLIP topography reliably excludes major motility disorders, patients could proceed with fundoplication without undergoing the additional burden of high resolution manometry (HRM) testing. Unfortunately, as of now, there are insufficient data available to justify a change in clinical practice. As a result, FLIP topography has remained relegated to a purely complimentary role.

To investigate this question, the investigators will perform FLIP topography (Endoflip 2.0) analysis on all patients undergoing routine evaluation for gastroesophageal reflux disease at the time of their pre-operative EGD. Those patients with repetitive antegrade contractions (RACs) on FLIP topography will be classified as having normal motility, while any other pattern will be considered abnormal. All patients will additionally complete a standard pre-operative reflux evaluation including HRM, Upper GI series (UGI), 48-hour wireless pH testing, and baseline GERD quality of life surveys. The investigators will then compare the results of the FLIP topography measurements to the results of the gold standard high-resolution manometry (HRM) in terms of the ability of the FLIP topography to differentiate between normal and impaired esophageal function in GERD patients. Subjects will then be followed through their anti-reflux operations and post-operative outcomes will be tracked with standardized symptom questionnaires at 1, 2 and 6 months post-operatively to evaluate for post-operative dysphagia and quality of life.

The investigators hypothesize that FLIP topography (Endoflip 2.0) in GERD patients will reliably identify individuals with normal motility, which will predict good outcomes after anti-reflux surgery. If this proves to be the case, formal high resolution manometry (HRM) testing would not be necessary prior to proceeding with fundoplication, allowing a paradigm shift in the pre-operative workup of this large population of patients.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or known history of GERD
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Previous esophageal or gastric surgery (including failed anti-reflux operation)
* Hiatal Hernia > 5cm based on upper GI
* Patients with a known major motility disorder (achalasia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who present to our comprehensive esophageal clinic for evaluation of suspected GERD meeting the inclusion/exclusion criteria will be asked to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2020-03-19 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Concordance between the presence of RACs versus the absence of major motility disorder | 6 months
  Evaluate the concordance between the presence of RACs on FLIP topography versus the absence of major motility disorder on HRM as defined by the Chicago classification system v3.

SECONDARY OUTCOMES:
Concordance between the presence of RACs versus distal esophageal amplitude | 6 months
  Evaluate the concordance between the presence of RACs on FLIP topography versus the finding of distal esophageal amplitude >20mmHg as a surrogate for adequate esophageal function for Nissen fundoplication.

OTHER OUTCOMES:
Evaluate patient satisfaction using study questionnaire | 6 months
  Evaluate patient satisfaction with the FLIP topography procedure compared to traditional High Resolution Manometry (HRM) testing using a questionnaire to rate pain, discomfort, and anxiety as "not at all", "a little", "some" or "a lot".
Post-Fundoplication Dysphagia | 6 months
  Assess rates of post-fundoplication dysphagia in patients with and without RACs on FLIP topography as determined by GERD-HRQL (gastroesophageal reflux disease health-related quality of life) scale.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No